CLINICAL TRIAL: NCT05421598
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Dose Ranging Study to Assess the Efficacy, Safety, and Tolerability of Subcutaneous Amlitelimab in Adult Participants With Moderate-to-severe Asthma
Brief Title: Dose Ranging Study of Amlitelimab in Adult Participants With Moderate-to-severe Asthma
Acronym: TIDE-asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRI17509; U1111-1272-2612 (Registry Identifier: ICTRP); 2024-510641-33 (Registry Identifier: CTIS); 2022-000065-41 (EudraCT Number)
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Amlitelimab dose level 1 (Experimental): Initial loading dose of amlitelimab on Day 1, followed by one injection of amlitelimab dose level 1 every 4 weeks (Q4W) until Week 20 (inclusive) and every 12 weeks (Q12W) starting from Week 24 and thereafter.
  Interventions: Drug: Amlitelimab
- Amlitelimab dose level 2 (Experimental): Initial loading dose of amlitelimab on Day 1, followed by one injection of amlitelimab dose level 2 Q4W until Week 20 (inclusive) and Q12W starting from Week 24 and thereafter.
  Interventions: Drug: Amlitelimab
- Amlitelimab dose level 3 (Experimental): Initial loading dose of amlitelimab on Day 1, followed by one injection of amlitelimab dose level 3 Q4W until Week 20 (inclusive) and Q12W starting from Week 24 and thereafter.
  Interventions: Drug: Amlitelimab
- Placebo (Placebo Comparator): Initial loading dose of amlitelimab matching placebo on Day 1, followed by one injection of amlitelimab matching placebo Q4W until Week 20 (inclusive) and Q12W starting from Week 24 and thereafter.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amlitelimab — Injection solution Subcutaneous injection
  Other Names: SAR445229
  Arms: Amlitelimab dose level 1; Amlitelimab dose level 2; Amlitelimab dose level 3
Drug: Placebo — Injection solution Subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a parallel, Phase 2, global, multicenter, randomized, double-blind, placebo-controlled, dose-ranging, four-arms study for treatment.

The purpose of this study is to assess the efficacy, safety, and tolerability of add-on therapy with amlitelimab in adult participants with moderate-to-severe asthma.

Study details include:

* The study duration (per participant) will be up to approximately 76 weeks for participants not going into LTS study and will be up to approximately 64 weeks for participants going into LTS study.
* The randomized treatment duration will be up to approximately 60 weeks.
* The scheduled number of visits will be 13.

ELIGIBILITY:
Inclusion Criteria:

* The participant must be between the ages of 18 and 75 inclusive at the time of signing the informed consent.
* Moderate to severe asthma diagnosed by a physician for ≥ 12 months according to stages 4 and 5 of the Global Initiative for Asthma (GINA ).
* Participants on existing therapy with medium to high doses of ICS (≥500 μg fluticasone propionate daily or comparable ICS dose in combination with at least one additional controller (e.g., long-acting beta agonist [LABA], leukotriene receptor antagonist [LTRA], long-acting muscarinic antagonist [LAMA], methylxanthines) for at least 3 months.
* ≥ 1 severe asthma exacerbation in the past year, with at least one exacerbation during treatment with medium to high doses of ICS (≥ 500 μg fluticasone propionate daily or one dose of ICS comparable).
* Participants with pre-BD forced expiratory volume in 1 second (FEV1) > 40% and < 80% of predicted normal at the screening visit.
* 5-item ACQ-5 score >1.5 at randomization.
* Participants with at least 12% reversibility and 200 mL post-BD FEV after administration of albuterol/salbutamol or levalbuterol/levosalbutamol at screening or documented history of a reversibility test.
* Weight ≥40 kg and ≤150 kg at the randomization visit.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Chronic lung disease other than asthma.
* Current or former smoker including active vaping of any products and/or marijuana with cessation within 6 months of screening or history of >10 pack-years.
* Participants who experience a deterioration of asthma that results in emergency treatment or hospitalization, or treatment with systemic steroids at any time from 1 month prior to screening.
* Suspicion of, or confirmed, coronavirus disease 2019 (COVID-19) infection during the screening period including known history of COVID-19 infection within 4 weeks prior to Screening; mechanical ventilation or extracorporeal membrane oxygenation (ECMO) secondary to COVID-19 within 3 months prior to Screening; COVID-19 infection who have not yet sufficiently recovered to participate in the procedures of a clinical trial.
* Active infection or history of clinically significant infection
* Known history of, or suspected, significant current immunosuppression, including history of invasive opportunistic or helminthic infections despite infection resolution or otherwise recurrent infections of abnormal frequency or prolonged duration.
* Active or latent tuberculosis (TB)
* A history of malignancy of any type (excluding basal and squamous cell skin cancer and in situ cervical carcinoma that has been excised and cured >3 years prior to baseline).
* History of solid organ transplant.
* Hepatitis B, C or HIV.
* Pregnant or breastfeeding.
* History (within last 2 years prior to Baseline) of prescription drug or substance abuse, including alcohol, considered significant by the Investigator.
* Any prior use of anti-OX40 or anti-OX40L mAb, including amlitelimab.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Annualized rate of severe exacerbation events over 48 weeks | Baseline through Week 48
  Severe exacerbation events are defined as: worsening of asthma requiring the use of systemic corticosteroids for ≥3 days or, in the case of a stable maintenance regimen of oral corticosteroids for the treatment of asthma, a doubling of the dose for 3 or more days; or hospitalization or emergency room visit because of asthma, requiring systemic corticosteroids.

SECONDARY OUTCOMES:
Change from baseline in pre-bronchodilator (BD) FEV1 at Week 48 | Baseline to Week 48
  Change from baseline in pre-bronchodilator (BD) FEV1 at Week 48.
Change from baseline in Asthma Control Questionnaire 5 (ACQ-5) score at Week 48 | Baseline to Week 48
  The ACQ-5 has five questions on the asthma symptoms. The score ranges from 0 (totally controlled) and 6 (severely uncontrolled). A high score indicates low asthma control.
Change from baseline in Asthma Quality of Life Questionnaire with Standardized Activities (AQLQ (S)) Self-Administered Score at Week 48 | Baseline to Week 48
  The AQLQ(S) is designed as a self-administered participant reported outcome to measure the functional impairments. The overall score is 1 to 7. Higher AQLQ scores indicate better health-related quality of life.
Change from baseline in post-BD FEV1 at Week 48 | Baseline to Week 48
  Change from baseline in post-BD FEV1 at Week 48.
The absolute change in the percent predicted FEV1 from baseline to Week 48 (pre-BD and post-BD) | Baseline to Week 48
  The absolute change in the percent predicted FEV1 from baseline to Week 48 (pre-BD and post-BD).
Change from baseline in ACQ-5 score at Weeks 2, 4, 8, 12, 24, 36, and 60 | Baseline to Weeks 2, 4, 8, 12, 24, 36, and 60
  The ACQ-5 has five questions on the asthma symptoms. The score ranges from 0 (totally controlled) and 6 (severely uncontrolled). A high score indicates low asthma control.
Time to first severe exacerbation event | Baseline through Week 48
  Severe exacerbation events are defined as: worsening of asthma requiring the use of systemic corticosteroids for ≥3 days or, in the case of a stable maintenance regimen of oral corticosteroids for the treatment of asthma, a doubling of the dose for 3 or more days; or hospitalization or emergency room visit because of asthma, requiring systemic corticosteroids.
Change from baseline in pre-BD and post-BD FEV1 | Baseline to Weeks 2, 4, 8, 12,16, 24, 36 and 60
  Change from baseline in pre-BD and post-BD FEV1.
Change from baseline in peak expiratory flow (PEF) and forced expiratory flow (FEF) 25-75% | Baseline to Weeks 4, 12, 24, 36, 48 and 60
  Change from baseline in peak expiratory flow (PEF) and forced expiratory flow (FEF) 25-75%.
Change from baseline in forced vital capacity (FVC) | Baseline to Weeks 4, 12, 24, 36, 48 and 60
  Change from baseline in forced vital capacity (FVC).
Change from baseline in FeNO at Weeks 2, 4, 8, 12, 16, 24, 36, 48 and 60 | Baseline to Weeks 2, 4, 8, 12, 16, 24, 36, 48 and 60
  Change from baseline in FeNO at Weeks 2, 4, 8, 12, 16, 24, 36, 48 and 60.
Annualized rate of loss of asthma control (LOAC) events during 48 weeks of treatment | Baseline through Week 48
  LOAC events are defined by one or several of the following criteria:
  A 30% or greater reduction from baseline in morning PEF on 2 consecutive days.
  ≥6 additional reliever puffs of short-acting beta-agonists (SABA) OR ≥4 additional puffs of low-dose inhaled corticosteroid (ICS)/formoterol in a 24-hour period (compared to baseline) on 2 consecutive days Increase in ICS ≥4 times than the Visit 2 dose Severe exacerbation event
Time to first LOAC event | Baseline through Week 48
  LOAC events are defined by one or several of the following criteria:
  A 30% or greater reduction from baseline in morning PEF on 2 consecutive days.
  ≥6 additional reliever puffs of short-acting beta-agonists (SABA) OR ≥4 additional puffs of low-dose ICS/formoterol in a 24-hour period (compared to baseline) on 2 consecutive days Increase in ICS ≥4 times than the Visit 2 dose Severe exacerbation event
Change from baseline in the Asthma Daytime Symptom Diary (ADSD) 7-item daily morning score and in the Asthma Nighttime Symptom Diary (ANSD) 7-item daily evening scores at Weeks 2, 4, 8, 12, 24, 36, 48, and 60 | Baseline to Weeks 2, 4, 8, 12, 24, 36, 48, and 60
  ADSD and ANSD have been designed to measure asthma symptoms. Both have overall score from 0- 10 with higher score indicating worse symptom.
Annualized rate of severe asthma exacerbations requiring hospitalization or emergency room or urgent care visit during 48 weeks of treatment | Baseline through Week 48
  Annualized rate of severe asthma exacerbations requiring hospitalization or emergency room or urgent care visit during 48 weeks of treatment.
Change from baseline in the numbers of inhalations/day of SABA or low-dose ICS/formoterol for symptom relief at Weeks 2, 4, 8, 12, 24, 36, 48, and 60 | Baseline to Weeks 2, 4, 8, 12, 24, 36, 48, and 60
  Change from baseline in the numbers of inhalations/day of SABA or low-dose ICS/formoterol for symptom relief at Weeks 2, 4, 8, 12, 24, 36, 48, and 60.
Serum amlitelimab concentrations measured throughout the study | Baseline thought Week 60
  Serum amlitelimab concentrations measured throughout the study.
Incidence of anti-amlitelimab antibody positive response | Baseline through Week 60
  Incidence of anti-amlitelimab antibody positive response.
Percentage of participants with treatment-emergent adverse events (TEAEs), including local reactions, AEs of special interest (AESIs), serious adverse events (SAEs) | Baseline through Week 60
  Percentage of participants with treatment-emergent adverse events (TEAEs), including local reactions, AEs of special interest (AESIs), serious adverse events (SAEs).
Incidence of potentially clinically significant laboratory test, vital signs, and ECG abnormalities in the treatment period | Baseline through Week 60
  Incidence of potentially clinically significant laboratory test, vital signs, and ECG abnormalities in the treatment period.
Change from baseline in Asthma Quality of Life Questionnaire with Standardized Activities (AQLQ (S)) Self-Administered Score at Weeks 2, 4, 8, 12, 24, 36, and 60 | Baseline to Weeks 2, 4, 8, 12, 24, 36, and 60
  The AQLQ(S) is designed as a self-administered participant reported outcome to measure the functional impairments. The overall score is 1 to 7. Higher AQLQ scores indicate better health-related quality of life.
Change from baseline in St. George's Respiratory Questionnaire (SGRQ) at Weeks 2, 4, 8, 12, 24, 36, 48, and 60 | Baseline to Weeks 2, 4, 8, 12, 24, 36, 48, and 60
  The SGRQ is designed to measure and quantify health status in adult patients with chronic airflow limitation. A global score ranges from 0 to 100 where 0 indicates best and 100 indicates worst health.
Proportion of participants with a decrease from baseline of at least 4 points in SGRQ total score at Week 48 | Week 48
  The SGRQ is designed to measure and quantify health status in adult patients with chronic airflow limitation. A global score ranges from 0 to 100 where 0 indicates best and 100 indicates worst health.
Change from baseline in ACQ-6 score and ACQ-7 at Weeks 2, 4, 8, 12, 24, 36, 48, and 60 | Baseline to Weeks 2, 4, 8, 12, 24, 36, 48, and 60
  The ACQ-6 is a validated asthma assessment tool that consists of 6 self-assessment questions. The overall scale ranges from 0 = 'totally controlled' to 6 = 'severely unc7ntrolled. The ACQ-7 is a validated asthma assessment tool that consists of 6 self-assessment questions. The overall scale ranges from 0 = 'totally controlled' to 6 = 'severely uncontrolled.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (113):
- United States (21):
  - University of California San Diego Health Site Number : 8400026, La Jolla, California
  - California Allergy and Asthma Medical Group, Inc. Site Number : 8400002, Los Angeles, California
  - Allergy Asthma Associates of Santa Clara Valley Site Number : 8400019, San Jose, California
  - Bensch Clinical Research LLC Site Number : 8400004, Stockton, California
  - Allianz Research Institute Site Number : 8400023, Westminster, California
  - Helix Biomedics, LLC Site Number : 8400029, Boynton Beach, Florida
  - Renaissance Research and Medical Group, Inc Site Number : 8400030, Cape Coral, Florida
  - Beautiful Minds Clinical Research Center Site Number : 8400027, Cutler Bay, Florida
  - Reliable Clinical Research, LLC Site Number : 8400020, Hialeah, Florida
  - Savin Medical Group, LLC Site Number : 8400015, Miami, Florida
  - Pines Care Research Center LLC Site Number : 8400028, Pembroke Pines, Florida
  - Treasure Valley Medical Research Site Number : 8400031, Boise, Idaho
  - The South Bend Clinic, LLC Site Number : 8400033, South Bend, Indiana
  - University of Kansas Medical Center Site Number : 8400016, Kansas City, Kansas
  - Johns Hopkins University School of Medicine Site Number : 8400012, Baltimore, Maryland
  - Headlands Research Detroit Site Number : 8400032, Southfield, Michigan
  - Henderson Clinical Trials Site Number : 8400037, Henderson, Nevada
  - Asthma and Allergy Center Site Number : 8400005, Toledo, Ohio
  - OK Clinical Research, LLC Site Number : 8400001, Edmond, Oklahoma
  - Allergy, Asthma and Clinical Research Center Site Number : 8400035, Oklahoma City, Oklahoma
  - TTS Research Site Number : 8400011, Boerne, Texas
- Argentina (9):
  - Investigational Site Number : 0320001, CABA, Buenos Aires
  - Investigational Site Number : 0320002, CABA, Buenos Aires
  - Investigational Site Number : 0320008, La Plata, Buenos Aires
  - Investigational Site Number : 0320009, Buenos Aires, Buenos Aires F.D.
  - Investigational Site Number : 0320006, Rosario, Santa Fe Province
  - Investigational Site Number : 0320007, Rosario, Santa Fe Province
  - Investigational Site Number : 0320005, Rosario, Santa Fe Province
  - Investigational Site Number : 0320004, Buenos Aires
  - Investigational Site Number : 0320003, Ciudad Autonoma Buenos Aires
- Brazil (8):
  - CEDOES - Centro de Diagnostico e Pesquisa de Osteoporose do ES Site Number : 0760002, Vitória, Espírito Santo
  - Proar Site Number : 0760004, Salvador, Estado de Bahia
  - Centro Avancado de Oncologia CECAN - Liga Contra o Cancer Site Number : 0760010, Natal, Rio Grande do Norte
  - Instituto Mederi de Pesquisa e Saude Site Number : 0760001, Passo Fundo, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericordia de Porto Alegre Site Number : 0760007, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS Site Number : 0760006, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas de Sao Paulo Site Number : 0760008, São Paulo, São Paulo
  - Clinica de Alergia Martti Antila Site Number : 0760003, Sorocaba, São Paulo
- Canada (5):
  - Investigational Site Number : 1240006, Brampton, Ontario
  - Investigational Site Number : 1240008, Ottawa, Ontario
  - Investigational Site Number : 1240005, Toronto, Ontario
  - Investigational Site Number : 1240007, Trois-Rivières, Quebec
  - Investigational Site Number : 1240003, Québec
- Chile (8):
  - Investigational Site Number : 1520006, Talca, Maule Region
  - Investigational Site Number : 1520007, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520009, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520008, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520005, Quillota, Región de Valparaíso
- Hungary (8):
  - Investigational Site Number : 3480007, Budapest
  - Investigational Site Number : 3480009, Edelény
  - Investigational Site Number : 3480011, Gödöllö
  - Investigational Site Number : 3480002, Hajdunánás
  - Investigational Site Number : 3480004, Mosonmagyaróvár
  - Investigational Site Number : 3480006, Püspökladány
  - Investigational Site Number : 3480012, Százhalombatta
  - Investigational Site Number : 3480003, Szombathely
- Italy (4):
  - Investigational Site Number : 3800002, Cona (FE), Emilia-Romagna
  - Investigational Site Number : 3800003, Rome, Lazio
  - Investigational Site Number : 3800004, Napoli
  - Investigational Site Number : 3800001, Verona
- Japan (17):
  - Investigational Site Number : 3920014, Narita-shi, Chiba
  - Investigational Site Number : 3920002, Kamakura-shi, Kanagawa
  - Investigational Site Number : 3920016, Yokohama, Kanagawa
  - Investigational Site Number : 3920006, Yokohama, Kanagawa
  - Investigational Site Number : 3920013, Nankoku-shi, Kochi
  - Investigational Site Number : 3920015, Kumamoto, Kumamoto
  - Investigational Site Number : 3920010, Sakai-shi, Osaka
  - Investigational Site Number : 3920017, Chuo-ku, Tokyo
  - Investigational Site Number : 3920005, Chuo-ku, Tokyo
  - Investigational Site Number : 3920004, Chuo-ku, Tokyo
  - Investigational Site Number : 3920020, Kiyose-shi, Tokyo
  - Investigational Site Number : 3920001, Shinagawa-ku, Tokyo
  - Investigational Site Number : 3920011, Shinjuku-ku, Tokyo
  - Investigational Site Number : 3920009, Tachikawa-shi, Tokyo
  - Investigational Site Number : 3920018, Toshima-ku, Tokyo
  - Investigational Site Number : 3920008, Fukuoka
  - Investigational Site Number : 3920019, Hiroshima
- Mexico (6):
  - Investigational Site Number : 4840001, Guadalajara, Jalisco
  - Investigational Site Number : 4840005, Guadalajara, Jalisco
  - Investigational Site Number : 4840002, Chihuahua City
  - Investigational Site Number : 4840004, Durango, Durango
  - Investigational Site Number : 4840006, Tlalnepantla
  - Investigational Site Number : 4840008, Yucatán
- Poland (6):
  - Investigational Site Number : 6160001, Poznan, Greater Poland Voivodeship
  - Investigational Site Number : 6160006, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number : 6160004, Bialystok, Podlaskie Voivodeship
  - Investigational Site Number : 6160003, Elblag
  - Investigational Site Number : 6160002, Gdansk
  - Investigational Site Number : 6160007, Tarnów
- South Africa (8):
  - Investigational Site Number : 7100007, Benoni
  - Investigational Site Number : 7100002, Cape Town
  - Investigational Site Number : 7100005, Cape Town
  - Investigational Site Number : 7100001, Cape Town
  - Investigational Site Number : 7100003, Durban
  - Investigational Site Number : 7100006, George
  - Investigational Site Number : 7100008, Johannesburg
  - Investigational Site Number : 7100004, Middelburg
- South Korea (7):
  - Investigational Site Number : 4100004, Daegu, Daegu
  - Investigational Site Number : 4100003, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100005, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100006, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100007, Seongnam-si, Gyeonggi-do
- Turkey (Türkiye) (5):
  - Investigational Site Number : 7920001, Istanbul
  - Investigational Site Number : 7920003, Izmir
  - Investigational Site Number : 7920008, Kayseri
  - Investigational Site Number : 7920005, Kocaeli
  - Investigational Site Number : 7920002, Mersin
- Investigational Site Number : 8260001, Bradford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: DRI17509 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25227&tenant=MT_SNY_9011